CLINICAL TRIAL: NCT04907409
Title: Home OCT Fluid Visualization Agreement Study at Multiple Retinal Clinics With Placement of One Home OCT Device in the Home of Each NV-AMD Subject in the US for 5 Weeks
Brief Title: Home OCT Fluid Visualization Agreement Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2021.001
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-01

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single arm study of home monitoring with the NVHO for 5 weeks with office visits at enrollment, Week 1 and Week 5 (Exit Visit) and, when applicable, Interim Visit(s) triggered by ongoing review by the Reading Center. The study will enroll subjects diagnosed with NV-AMD in at least one eye with attention to the proportion of eyes with IRF and/or SRF. The enrolled eligible subjects will be instructed to self-image the study eye(s) once daily for 5 weeks using a NVHO device at home with scheduled in-office examinations at Week 1, Week 5 and Interim Visits, when applicable, with additional in-office Cirrus volume scans acquired at these office visits. The self-imaging data on the NVHO will be automatically uploaded to the Notal Health Cloud and from there the reconstructed volume scans will sent to the study database.

DETAILED DESCRIPTION:
The objectives of this study are to (1) evaluate the agreement, via positive percent agreement (PPA) and negative percent agreement (NPA), between OCT images captured by the NVHO and by the Zeiss Cirrus HD-OCT in the visualization of fluid as identified by a RC, in the central 10 degrees of the macula of NV-AMD patients, and (2) evaluate the ability of subjects diagnosed with NV-AMD to set up the device and self-image their eyes at home with the NVHO device (rate of successful imaging attempts).Description of Study Visits and Procedures:

Enrollment Visit:

At this visit, the exams will be conducted in the following order:

1. Subject will be informed concerning the study and sign the Informed Consent Form (ICF) prior to the conduct of any study procedures.
2. The following data will be collected for each study subject:

   1. Subject's date of birth (DOB) (if allowed) or age
   2. Gender
   3. Race
   4. Ethnicity
   5. Level of education
3. Eye exams, including Snellen BCVA and subjective symptoms (visual distortions, blurry vision, and scotoma), will be performed on both eyes on the day of the visit.
4. Both eyes of the subject will be imaged using a commercial Zeiss Cirrus OCT using the 6mm X 6mm, 512 X 128 volume scan program, with a maximum of three attempts for each eye to reach an acceptable image quality per the Cirrus User's Guide and reviewed by the PI to determine fluid status.
5. One or both eye(s) of the subject that meets all screening criteria, including having a diagnosis of NV-AMD in at least one eye previously or at the enrolment visit, will be enrolled in the study.

   * Subjects who do not meet all screening criteria will be deemed a screen failure and will be exited from the study.
   * Study eyes enrolled with fluid in the primary study eye, may receive treatment during the Week 1 Visit.
   * If in the investigator's opinion, the treatment cannot be delayed by approximately 7 days until the Week 1 visit, the subject will be exited from the study as a Screen Failure.

   NOTE: For the subjects with both eyes with NV-AMD, one eye will be randomly selected as the primary eye during enrollment and the other will be the secondary eye. For subjects with only one eye with NV-AMD, the fellow eye with dry AMD may be enrolled. For such subjects, the NV-AMD eye will be the primary eye and the other eye will be the secondary eye.
6. The following data will be collected for the study eye:

   1. Qualifying diagnosis for the study eye from the subject's medical record
   2. From the subject's medical record, the presence of other ophthalmic conditions including but not limited to:

   i. Cataract ii. Glaucoma iii. Dry Eye iv. Other macula findings
7. The subject will receive a general overview (including a description of the device and a review of the NVHO set-up guide) of the self-operation of the NVHO device at the investigational clinic facility by trained study personnel.
8. The subject will be (1) reminded that the NVHO device will be delivered to their home and (2) instructed to self-image the study eye(s) once daily using a NVHO device at home for 5 weeks and the Week 1 and Week 5 visits will be scheduled.
9. Collect AEs, if applicable.

Home Set-up with Remote Assistance (NVHO Setup Period)

Following confirmation of subject eligibility at the Enrollment Visit and the subject is enrolled in the study:

1. The subject will be contacted by the NVDC to verify their delivery address.
2. The device will be delivered to the subject's home, with confirmation sent back to the NVDC.
3. Remote support is available by the Notal Vision Diagnostic Clinic (NVDC) via phone during normal business hours, if needed.
4. The subject will follow the steps detailed in the Set-up Guide included in the box. This is considered NVHO Setup Period.

   Note: A care giver, family member or friend is allowed to assist. At most four additional calibrations can be performed, on the same day or different consecutive days, for each study eye if the calibration is not successful.

   Note: If an eye cannot calibrate during 5 separate attempts, the subject will be notified by the NVDC to discontinue self-imaging this eye and NVDC will collect the corresponding information such as the corresponding eye, self-image discontinuation reason, and the self-image stopping date. If there is a fellow eye also enrolled in the study, the fellow eye will continue.
5. Collect AEs, if applicable.

In-Home Phase (Day 1 to Day 35 post NVHO Setup Period) Following set-up of the NVHO,

1. Day 1: The subject will perform the first self-imaging session with the NVHO device on both eyes followed by automated transmission of the scans. This first session will be considered a practice session.
2. Days 2-35: The subject will perform one self-imaging session each day on the study eye(s) with the NVHO device followed by automated transmission. Each scan has a reliability score provided by the NVHO.

   Note: If an eye fails to self-image five consecutive times, the subject will be notified by the NVDC to discontinue self-imaging this eye and NVDC will collect the corresponding information such as the corresponding eye, self-image discontinuation reason, and the self-image stopping date. If there is a fellow eye also enrolled in the study, the fellow eye will continue.
3. Collect AEs, if applicable, as reported by telephone call or office visit to the investigational site.

Week 1 (Post NVHO Setup Period)

Subjects will return to the clinic for an office visit one week after the NVHO Setup Period (Home Set-up). The sponsor will provide transportation upon request. At this visit, the exams will be conducted in the following order:

1. Eye exams, including Snellen BCVA and subjective symptoms (visual distortions, blurry vision, and scotoma) will be performed on both eyes on the day of the visit.
2. Both eyes of the subject will be imaged using a commercial Zeiss Cirrus OCT using the 6mmX6mm, 512X128 volume scan program, with a maximum of three attempts for each eye to reach an acceptable image quality per the Cirrus User's Guide and reviewed by the PI to determine fluid status.
3. Initiate standard of care and treatment, if necessary.
4. Collect AEs, if applicable. Week 5 / Exit (Post NVHO Setup Period)

Subjects will return to the clinic for an office visit five weeks after the NVHO Setup Period (Home Set-up). At this visit, the exams will be conducted in the following order:

1. Eye exams, including Snellen BCVA and subjective symptoms (visual distortions, blurry vision, and scotoma) will be performed on both eyes on the day of the visit.
2. Both eyes of the subject will be imaged using a commercial Zeiss Cirrus OCT using the 6mmX6mm, 512X128 volume scan program, with a maximum of three attempts for each eye to reach an acceptable image quality per the Cirrus User's Guide and reviewed by the PI to determine fluid status.
3. Initiate standard of care and treatment, if necessary.
4. Collect AEs, if applicable.
5. Exit subject from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the ability to speak, read and understand English.
2. Ability to understand and agree to contents of informed consent either in writing or verbally.
3. Age 55 or older at the Enrollment Visit.
4. Adults diagnosed with NV-AMD in at least one eye based on the subject's medical record. Fellow eyes diagnosed with dry AMD may be included as secondary eyes to a primary eye diagnosed with NV-AMD.

   Note: eyes whit other pathologies including pseudocysts, outer retinal tabulations, pigments epithelial, detachments, hemorrhage, sub retinal hyper reflective material (SHRM), geographic atrophy and sub RPE, hypo reflective areas can be enrolled.
5. Best corrected Visual Acuity of 20/320 or better in eyes that will perform self-imaging.
6. Available and willing to set up a device and conduct self-imaging at their home.

Exclusion Criteria:

1. Anti-VEGF treatment for NV-AMD in the study eye(s) at the screening visit.
2. Any other retinal disease requiring steroidal or anti-VEGF injections.
3. Prior experience with the NVHO device.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects diagnosed with neovascular age-related macular degeneration (NV-AMD) in at least one eye at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Positive percent agreement | 1 month following reading center grading completion
  Positive percent agreement (PPA) of fluid status when comparing the fluid status in the central 3mm X 3mm of the NVHO volume scan graded by an independent reading center to the fluid status in the central 3mm X 3mm of Cirrus volume scan graded by an independent reading center.
Negative percent agreement | 1 month following reading center grading completion
  Negative percent agreement (NPA) of fluid status when comparing the fluid status in the central 3mm X 3mm of the NVHO volume scan graded by an independent reading center to the fluid status in the central 3mm X 3mm Cirrus volume scan graded by an independent reading center.
Percentage of subjects who successfully completed the setup of the NVHO device | 5-10 minutes
  Percentage of subjects who successfully completed the setup of the NVHO, indicated by the initiation of the tutorial.
Percentage of subjects who Successful completed NVHO self-imaging | 2-3 minutes
  Percentage of subjects who Successful completed NVHO self-imaging, namely a volume macular scan has been captured.

SECONDARY OUTCOMES:
Percentage of all sessions that were transmission successfully | 10-15 minutes
  Percentage of sessions transmitted successfully to the Notal Health Cloud to the Notal Health Cloud .
Percentage of sessions containing self-imaging that were transmitted successfully | 10-15 minutes
  Percentage of sessions containing self-imaging that were transmitted successfully to the Notal Health Cloud.

CONTACTS AND LOCATIONS:
Overall Officials: Gidi Benyamini, MD, Study Director — Druyanov 5, Tel Aviv Israel
Locations (7):
- United States (7):
  - Georgia Retina, Marietta, Georgia
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Elman Retina Group, P.A., Glen Burnie, Maryland
  - Ophthalmic Cons. of Boston, Boston, Massachusetts
  - Pepose Vision Institute/Midwest Vision Research Foundation, Chesterfield, Missouri
  - Wagner Macula & Retina Center, Norfolk, Virginia
  - Virginia Eye Institute, Richmond, Virginia